CLINICAL TRIAL: NCT05247619
Title: A Clinical Study to Explore the Efficacy and Safety of Tislelizumab in Combination With Bevacizumab and Chemotherapy in Patients With Persistent, Recurrent, or Metastatic Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Jianqing Zhu, MD, Chief physician, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-2007
Record Dates: First submitted 2022-01-24; First posted 2022-02-21 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — tislelizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Tislelizumab + Bevacizumab + Paclitaxel + Cisplatin/Carboplatin
  Interventions: Drug: Tislelizumab / Bevacizumab/Paclitaxel/Cisplatin/Carboplatin

INTERVENTIONS:
Drug: Tislelizumab / Bevacizumab/Paclitaxel/Cisplatin/Carboplatin — Tisleliumab 200mg, Bevacizumab 7.5mg/kg, Paclitaxel 175mg/m2, and Cisplatin 50mg/m2 (or Carboplatin AUC5) IV on day 1 of every 21-day cycle.

SUMMARY:
Efficacy and safety of Tislelizumab combined with Bevacizumab and chemotherapy in patients with persistent, recurrent or metastatic cervical cancer.

DETAILED DESCRIPTION:
The current standard treatment for persistent, metastatic and recurrent cervical cancer is platinum-based combination chemotherapy as its first-line treatment option. However, the current treatment plan still can not meet the clinical needs of cervical cancer treatment, most patients will progress about 6 months after first-line treatment.

At present, there are many clinical research evidence to support the PD-1 antibody for the treatment of recurrent cervical cancer. Immunotherapy can restore the environment of immune support and promote vascular normalization, while anti-angiogenesis can not only normalize tumor vessels, but also block immunosuppressive signals through many ways, so the two mechanisms complement each other. Inhibition of these two pathways will bring better and more lasting clinical benefits to cervical cancer patients.

This study explores the efficacy and safety of tirelizumab combined with bevacizumab and chemotherapy in patients with persistent, recurrent, or metastatic cervical cancer. combining with immune checkpoint inhibitors on the basis of standard treatment regimens has a more potent and durable antitumor ability mechanistically, no significant adverse reactions overlap between immunotherapy and existing standard regimens from a safety perspective, and multiple immune checkpoint combined with antiangiogenic studies confirm safety in cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and signature of informed consent;
2. Age ≥18;
3. Eastern United States Cancer Collaboration Group (ECOG) score 0-1;
4. Patients with metastatic (IVB), persistent or first recurrent cervical cancer is unsuitable for surgical treatment;
5. Histopathology was defined as: cervical squamous cell carcinoma, adenocarcinoma, adenosquamous carcinoma, patients included in adenocarcinoma histology will be limited to 20% of the entire study population;
6. Patients must have lesions that can be measured according to RECIST v1.1 criteria;
7. The main organs function well and are defined as:

   * Patients received no blood, platelet transfusion or growth factor support treatment within 14 days ≤ the beginning of treatment and was required to:

     * x 109/L ANC ≥1.5
     * Platelet ≥100 x 109/L
     * g/L ≥90
   * AST and ALT≤2.5 times ULN (5 times if liver metastasis occurs)
   * Serum total bilirubin ≤ ULN 1.5 times
   * Serum creatinine <1.5x upper limit (ULN)
   * Urine routine examination, urine protein <2+
   * The internationally standardized ratio (INR)≤1.5 or prothrombin time ULN 1.5 times
   * The activated partial thromboplastin time (aPTT)≤1.5 times ULN time
   * Serum albumin ≥30 g/L
8. Life expectancy ≥3 months;
9. Pregnant women must agree to effective contraception ≥120 days during the study period and after the last drug administration, and the results of serum pregnancy tests were negative 7 days ≤ before the first drug administration;

Exclusion Criteria:

1. Patients whose bilateral hydronephrosis can not be alleviated by ureteral stent or percutaneous drainage; non-communicable cystitis CTCAE(5.0 Edition)≥ grade 2;
2. Exclusion criteria of bevacizumab, i.e. clinical significance of cardiovascular and cerebrovascular diseases, abdominal fistula or gastrointestinal perforation history, acute intestinal obstruction or subimpedance, active bleeding;
3. hypertension (systolic blood pressure greater than 140 mmHg and/or diastolic blood pressure greater than 90 mmHg), hypertension crisis or history of hypertensive encephalopathy, which remains uncontrolled under medication;
4. Previous medical history showing newly discovered thrombotic disease within 6 months of screening or during screening; patients with severe wound nonunion, ulcers or fractures;
5. Patients with other malignancies and brain metastases;
6. Patients with central nervous system diseases, including uncontrolled seizure standard drug therapy, or historical cerebrovascular accidents (CVA, stroke), transient ischemic attacks (TIA) or subarachnoid hemorrhage within six months.
7. Previous treatment with antiprogrammed cell death protein-1(anti PD-1), antiprogrammed death ligand-1(anti PD-L1) or anti PD-L2 drugs, or have received another drug treatment (e.g., cytotoxic T lymphocyte-associated antigen-4[ CTLA-4]、OX-40,] antigen patients CD137[ tumor necrosis factor receptor superfamily member 9(TNFRSF9)]; A patient who has previously received any VEGF drugs, including bevacizumab.
8. Patients who received live vaccinations or had undergone major surgery within 30 days prior to the first administration of the study; patients who were expected to undergo invasive surgery during treatment;
9. Active autoimmune diseases requiring systemic treatment in the past two years;
10. ≤14 days before the first administration of the study drug, any condition requiring systemic treatment with corticosteroids (prednisone or equivalent >10 mg/ days) or other immunosuppressive drugs;
11. History of known human immunodeficiency virus (HIV) infection;
12. Untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers (HBV DNA >500 IU/mL) or active HCV carriers with detectable levels; Note: Non-active hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B patients (HBV DNA <500 IU/mL) can be enrolled;
13. History of interstitial lung disease, non-infectious pneumonia or uncontrolled disease, including pulmonary fibrosis, acute lung disease, etc;
14. Severe chronic or active infections (including tuberculosis infections) requiring systemic antimicrobial, antifungal or antiviral therapy within 14 days prior to the first administration of the study drug Note: Patients with viral hepatitis are allowed antiviral therapy;
15. with severe cardiovascular diseases such as myocardial infarction, acute coronary syndrome, or coronary angioplasty/stenting/bypass transplantation in the past 6 months, or new york heart disease association (NYHA) class ii-class IV congestive heart failure (CHF), or history of class NYHA III or IV CHF;
16. who are known to be allergic to components of a study drug or its analog;
17. Participate in another clinical study at the same time, unless it is an observational (non-intervention) clinical study or at a follow-up period of an intervention study;
18. Pregnant or lactating women;
19. Previous heterogenous stem cell transplantation or organ transplantation;
20. Other conditions judged by the researchers did not meet the requirements of the group.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
mPFS | The time from the first dosing of the study drug until the first objective recording of disease progression or death from any cause, whichever occurred first, up to approximately 24 months.
  mPFS of Tislelizumab in combination with bevacizumab and chemotherapy in patients with persistent, relapsed, or metastatic cervical cancer was assessed by investigators according to RECIST v1.1

SECONDARY OUTCOMES:
ORR | Up to approximately 24 months
  ORR of Tislelizumab in combination with bevacizumab and chemotherapy in patients with persistent, relapsed, or metastatic cervical cancer were assessed by investigators according to RECIST v 1.1
DCR | Up to approximately 24 months
  DCR of Tislelizumab in combination with bevacizumab and chemotherapy in patients with persistent, relapsed, or metastatic cervical cancer was assessed by investigators according to RECIST v1.1
DOR | DOR: refers to the time from the beginning of the first assessment of a tumor as CR or PR to the first assessment of PD or death from any cause, up to 24 months.
  DOR of Tislelizumab in combination with bevacizumab and chemotherapy in patients with persistent, relapsed, or metastatic cervical cancer were assessed by investigators according to RECIST v 1.1
Adverse Event (AE) | The time from the first dosing of the study drug until 90 days after last dose of study treatment (Up to approximately 27 months )
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be presented.
Serious AE (SAE) | The time from the first dosing of the study drug until 90 days after last dose of study treatment (Up to approximately 27 months )
  An SAE is defined as any untoward medical occurrence that, at any dose: a.) Results in death; b.) Is life-threatening; c.) Requires inpatient hospitalization or prolongation of existing hospitalization; d.) Results in persistent or significant disability/incapacity; e.) Is a congenital anomaly/birth defect; f.) Other important medical events; h.) Is a new cancer (that is not a condition of the study) or i.) Is associated with an overdose. The number of participants who experience an SAE will be presented.
Immune-related AE (irAE) | The time from the first dosing of the study drug until 90 days after last dose of study treatment (Up to approximately 27 months )
  AEs associated with tislelizumab exposure may be a result of an immune response. These irAEs may occur shortly after the first dose or several months after the last dose of tislelizumab treatment .

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China